CLINICAL TRIAL: NCT07057557
Title: Comparison of Postoperative Pain After Application of Aloe Vera Gel Dressings With Conventional Paraffin-Based Tulle Dressings at Split-Thickness Skin Graft Donor Site
Brief Title: Aloe Vera vs Paraffin Tulle Dressings for Pain Management in Split Thickness Skin Graft Donor Sites
Acronym: AloePaTu
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King Edward Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 396/RC/KEMU
Record Dates: First submitted 2025-06-30; First posted 2025-07-10 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Skin Graft Wounds; Donor Site Complication; Pain, Postoperative; Skin Transplantation
MeSH Terms: conditions — Pain, Postoperative | interventions — aloe vera gel extract hydrogel dressing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aloe Vera Gel Dressing (Experimental): Participants in this group will receive Aloe Vera gel applied directly to the split-thickness skin graft donor site
  Interventions: Other: Aloe Vera Gel Dressing
- Paraffin-Based Tulle Dressing (Conventional Dressing) (Active Comparator): Participants in this group will receive standard paraffin-based tulle dressing with chlorhexidine on the donor site.
  Interventions: Other: Paraffin-Based Tulle Dressing

INTERVENTIONS:
Other: Aloe Vera Gel Dressing — Participants in this arm will receive Aloe Vera gel applied directly to the split-thickness skin graft (STSG) donor site immediately after graft harvesting. The Aloe Vera gel will be applied in a sterile manner, followed by secondary dressing with dry gauze and crepe bandage. Pain will be assessed on postoperative day 7 using the Visual Analogue Scale (VAS).
  Arms: Aloe Vera Gel Dressing
Other: Paraffin-Based Tulle Dressing — Participants in this arm will receive a conventional paraffin-based tulle dressing impregnated with chlorhexidine applied to the STSG donor site. The dressing will be followed by secondary coverage with dry gauze and crepe bandage. Pain will be assessed on postoperative day 7 using the Visual Analogue Scale (VAS).
  Arms: Paraffin-Based Tulle Dressing (Conventional Dressing)

SUMMARY:
The goal of this clinical trial is to learn if Aloe Vera gel dressing helps reduce pain better than traditional paraffin-based tulle dressing at the donor site of split-thickness skin grafts in adult patients aged 18 to 60. The main questions it aims to answer are:

Does Aloe Vera gel dressing reduce postoperative pain more effectively than paraffin-based tulle dressing on the 7th day after surgery?

Is there a difference in the need for additional pain medication between the two groups?

Researchers will compare Aloe Vera gel dressing to paraffin-based tulle dressing to see if Aloe Vera leads to better pain control.

Participants will:

Undergo split-thickness skin graft surgery

Receive either Aloe Vera gel dressing or paraffin-based tulle dressing at the donor site

Have pain measured using a visual analogue scale (VAS) on the 7th day after surgery

Be given pain medication if their pain score is 4 or higher, and the amount used will be recorded

DETAILED DESCRIPTION:
This randomized controlled trial aims to evaluate the effectiveness of Aloe Vera gel dressings compared to conventional paraffin-based tulle dressings in reducing postoperative pain at the donor site of split-thickness skin grafts (STSG). The study will be conducted in the Department of Plastic Surgery, Mayo Hospital, Lahore, over a period of six months.

Split-thickness skin grafting is a common reconstructive surgical procedure. Although effective, it creates a donor site wound that often causes significant postoperative pain, potentially affecting patient recovery and satisfaction. While paraffin-based tulle dressings are widely used, they may not offer optimal pain relief. Aloe Vera gel, due to its anti-inflammatory, analgesic, and wound-healing properties, is a promising alternative that has shown benefit in burn wounds and other superficial skin injuries.

A total of 72 patients (aged 18-60 years, of either gender) requiring STSG will be enrolled and randomized into two equal groups:

Group A will receive Aloe Vera gel dressings applied directly to the donor site.

Group B will receive conventional paraffin-based tulle dressings.

Both groups will undergo secondary dressing using dry gauze and crepe bandages. All procedures will be performed under general anesthesia, and grafts will be harvested at a uniform thickness (0.25-0.30 mm) using an electric dermatome.

Pain will be assessed using the Visual Analogue Scale (VAS) on postoperative day 7. Analgesic use (specifically nalbuphine) will be recorded for patients reporting a VAS score ≥4. The primary outcome is the difference in mean pain scores between the two groups; secondary data includes the total analgesic consumption.

This study will provide evidence on whether Aloe Vera gel dressing is a more effective alternative to conventional dressing in managing donor site pain following skin grafting, potentially improving patient outcomes and influencing future dressing protocols.

ELIGIBILITY:
Inclusion Criteria:

* • Patients aged 18-60 years of age of either gender needing Split thickness skin graft

Exclusion Criteria:

* • Patients known to have exaggerated/diminished pain response due to certain medical conditions (e.g. diabetes, neuropathy, chemotherapy, opioids etc.)

  * Patients allergic to either dressings

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-08-05 (Actual); Primary Completion 2026-02-05 (Estimated); Study Completion 2026-04-14 (Estimated)

PRIMARY OUTCOMES:
Pain Score at Donor Site on Postoperative Day 7 | 7 days after surgery
  Postoperative pain will be measured using the Visual Analogue Scale (VAS), which ranges from 0 (no pain) to 10 (worst possible pain).

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Hospital Lahore, Lahore, Punjab Province, Pakistan